CLINICAL TRIAL: NCT01933815
Title: Phase 1/2 Dose-Escalation Study of TPI 287 in Combination With Bevacizumab Followed by Randomized Study of the Maximum Tolerated Dose of TPI 287 in Combination With Bevacizumab Versus Bevacizumab Alone in Adults With Recurrent Glioblastoma
Brief Title: Dose-Escalation Study of TPI 287 + Avastin Followed by Randomized Study of the Same Versus Avastin for Glioblastoma
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPI-287-17
Record Dates: First submitted 2013-08-26; First posted 2013-09-02 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2022-07

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma multiforme; Glioblastoma; Radiotherapy; Temozolomide; TPI 287; Taxoid; Avastin; Bevacizumab
MeSH Terms: conditions — Glioblastoma | interventions — TPI-287; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TPI 287 + bevacizumab (Experimental): All subjects in phase 1 & subjects randomized to the TPI 287 + bevacizumab arm in phase 2 will be administered a 1-hour IV infusion of TPI 287 once every 3 weeks (Days 1 & 22 of 42-day cycle) & a 30-90 minute IV infusion of bevacizumab once every 2 weeks (Days 1, 15, & 29).
  In phase 1, the dose of TPI 287 will be escalated in sequential dose cohorts of 3 to 6, while the dose of bevacizumab remains constant (10 mg/kg). The first 5 dose levels will be 140, 150, 160, 170, & 180 mg/m2. Dose levels beyond 180 mg/m2 will be increased in increments of 20 mg/m2. Three subjects will be treated at a dose level halfway between the dose level that exceeds the MTD and the dose level immediately prior to further refine the MTD.
  In phase 2, the dose of TPI 287 will be the MTD determined in phase 1, & the dose of bevacizumab will be the same as phase 1 (10 mg/kg).
  Subjects may continue on treatment unless they meet one or more of the protocol discontinuation criteria.
  Interventions: Drug: TPI 287; Drug: Bevacizumab
- Bevacizumab (Active Comparator): All subjects randomized to the bevacizumab alone arm in phase 2 will be administered bevacizumab as a 30 to 90 minute IV infusion once every 2 weeks (Days 1, 15, and 29 of a 42-day cycle). The dose of bevacizumab will be 10 mg/kg.
  Subjects will be withdrawn from the study if they meet one or more of the discontinuation criteria outlined in the protocol; however, treatment with bevacizumab may continue under the FDA approved labeling for bevacizumab at the discretion of the subject's doctor.
  All subjects in phase 1 will be administered TPI 287 in combination with bevacizumab (i.e., there will be no bevacizumab alone arm during phase 1).
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: TPI 287 — TPI 287 is a microtubule inhibitor belonging to the taxane diterpenoid (taxoid) family, and specifically to the abeotaxane class. TPI 287 is an Investigational Drug.
  Other Names: TPI-287; NBT 287
  Arms: TPI 287 + bevacizumab
Drug: Bevacizumab — Avastin (bevacizumab) is an FDA approved drug indicated for multiple cancers, including as a single agent for GBM for adult patients with progressive disease following prior therapy. Single agent effectiveness is based on improvement in objective response rate; no data is available demonstrating improvement in disease-related symptoms or survival with bevacizumab.
  Other Names: Avastin

SUMMARY:
This trial is divided into two parts, a dose-escalation study (phase 1) and a randomized study (phase 2).

The purpose of the dose-escalation study (phase 1) is to determine the safety, maximum tolerated dose (MTD), and efficacy of TPI 287 in combination with Avastin (bevacizumab) in subjects who have glioblastoma multiforme (GBM) that has progressed following prior radiation therapy and temozolomide (TMZ).

The purpose of the randomized study (phase 2) is to determine the safety and efficacy of the phase 1 MTD of TPI 287 in combination with bevacizumab versus bevacizumab alone in subjects who have GBM that has progressed following prior radiation therapy and TMZ.

DETAILED DESCRIPTION:
This multi-center trial is a phase 1/2 study that will be conducted in two sequential phases, phase 1 and phase 2.

Phase 1 of the trial is a dose-escalation study of the safety, tolerability (MTD), and efficacy of TPI 287 in combination with bevacizumab in subjects who have GBM that has progressed following prior radiation therapy and TMZ.

* All subjects will be administered TPI 287 as an intravenous (IV) infusion (target duration of 1 hour) once every 3 weeks (Days 1 and 22 of a 42-day cycle) and bevacizumab as a 30 to 90 minute IV infusion once every 2 weeks (Days 1, 15, and 29 of the 42-day cycle). The subsequent cycle will start 3 weeks after the last TPI 287 infusion and 2 weeks after the last bevacizumab infusion, maintaining the once every 3 week and once every 2 week schedule, respectively.
* The dose of TPI 287 will be escalated in sequential dose cohorts of 3 to 6 subjects, while the dose of bevacizumab remains constant (10 mg/kg). The initial cohort of 3 subjects will be treated at a TPI 287 dose of 140 mg/m2. The next four dose levels will be 150, 160, 170, and 180 mg/m2. Dose levels beyond 180 mg/m2 will be increased in increments of 20 mg/m2 (i.e., 200, 220, 240 mg/m2, etc.).
* Once a dose level is identified that exceeds the MTD, dose de-escalation will be used to further refine the MTD. Specifically, 3 subjects will be treated at an intermediate dose level, halfway between the dose level that exceeded the MTD and the dose level immediately prior (e.g., 230 mg/m2, if 240 mg/m2 exceeded the MTD).
* Subjects will be assigned to dose cohorts in the order that they are enrolled; there is no randomization for phase 1. Approximately 20 to 32 subjects are planned for enrollment in phase 1, depending on the dose level at which dose limiting toxicities (DLTs) are observed.
* Dose modifications and delays will be required as described in the protocol. Subjects may continue on treatment unless they meet one or more of the discontinuation criteria outlined in the protocol. Subjects who are discontinued prior to completing Cycle 1 for any reason other than toxicity will be replaced.
* Adverse events (AEs) and concomitant medications will be monitored throughout the study. Subjects will be given a diary to record any AEs or concomitant medications taken between visits. Additional safety evaluations will include physical examination (including neurologic examination), Karnofsky performance status (KPS), weight (body surface area, BSA), vital signs, hematology, serum chemistry, and urinalysis.
* Efficacy evaluations will include magnetic resonance imaging [MRI, including both pre and post-gadolinium T1-weighted scans and T2/fluid attenuated inversion recovery (FLAIR) images], corticosteroid usage, and neurologic status (as measured by neurologic exam and KPS).

Phase 2 of the trial is a randomized study of the safety and efficacy of the phase 1 MTD of TPI 287 in combination with bevacizumab versus bevacizumab alone in subjects who have GBM that has progressed following prior radiation therapy and TMZ.

* Sixty subjects will be randomized 1:1 to receive either TPI 287 in combination with bevacizumab or bevacizumab alone.
* For the combination arm, the subjects will be administered TPI 287 as an IV infusion (target duration of 1 hour) once every 3 weeks (Days 1 and 22 of a 42-day cycle) and bevacizumab as a 30 to 90 minute IV infusion once every 2 weeks (Days 1, 15, and 29 of the 42-day cycle). The dose of TPI 287 will be the MTD determined in phase 1, and the dose of bevacizumab will be the same as phase 1 (10 mg/kg).
* Subjects randomized to the bevacizumab alone arm will be administered 10 mg/kg bevacizumab as a 30 to 90 minute IV infusion once every 2 weeks (Days 1, 15, and 29 of the 42-day cycle).
* The same dose modifications and delays required in phase 1 will apply to phase 2. Subjects may continue on treatment unless they meet one or more of the discontinuation criteria outlined in the protocol. There will be no subject replacement for phase 2 of the trial.
* The safety and efficacy evaluations during phase 2 will be the same as those in phase 1. In addition, subjects participating in phase 2 will be telephoned every two months following the final study visit (4 weeks after the last dose of study drug) for up to two years after randomization to follow survival.
* Subjects that participate in phase 1 of the trial will not be eligible to participate in phase 2 of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven GBM
2. Disease progression following radiation and TMZ
3. Up to 2 prior relapses allowed
4. Baseline MRI within 17 days of Day 1 & on steroid dosage that has been stable or decreasing for at least 5 days
5. Recent resection of recurrent or progressive tumor allowed as long as at least 4 weeks have elapsed from date of surgery and the subject has recovered from surgery
6. Life expectancy >12 weeks
7. Eighteen years old or older
8. KPS equal to or greater than 70
9. Recovered from toxic effects of prior therapy to < Grade 2 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) prior to Day 1. Minimum duration required between prior therapy and Day 1 is:

   1. At least 12 weeks from completion of radiation therapy except if there is unequivocal evidence for tumor recurrence in which case at least 4 weeks
   2. 4 weeks from prior cytotoxic therapy
   3. 4 weeks from prior experimental drug
   4. 6 weeks from nitrosoureas
   5. 3 weeks from procarbazine
   6. 1 week for non-cytotoxic agents, such as interferon, tamoxifen, & cis-retinoic acid
10. Adequate bone marrow function (absolute neutrophil count > 1,500/mm3 and platelet count of > 100,000/mm3), adequate liver function [ALT and AST <3 x upper limit normal (ULN), alkaline phosphatase <2 x ULN, and total bilirubin <1.5 mg/dL], & adequate renal function (BUN and creatinine <1.5 x ULN)
11. Minimum hemoglobin of 9 g/dL
12. Males & women of childbearing potential must agree to abstain from sex or use an adequate method of contraception for the duration of study, & for 6 months after last dose of study drug
13. Signed & dated informed consent prior to Screening evaluations

Exclusion Criteria:

1. Radiographic evidence of contrast-enhancing tumor crossing midline, leptomeningeal dissemination, gliomatosis cerebri or infratentorial tumor
2. Evidence or suspicion of disease metastatic to sites remote from the supratentorial brain
3. Prior treatment with bevacizumab or other anti-vascular endothelial growth factor (VEGF) drugs
4. Prior treatment with tyrosine-kinase inhibitors targeting VEGF, platelet-derived growth factor, fibroblast growth factor, tyrosine kinase with immunoglobulin-like and epidermal growth factor-like domains 2 (TIE-2), or angiopoietin (or their receptors)
5. Prior treatment with histone deacetylase inhibitors or mammalian target of rapamycin (mTOR) inhibitors
6. Prior treatment with TPI 287
7. Treatment with Enzyme-Inducing Anti-Epileptic Drugs within 2 weeks prior to Day 1
8. Treatment with drugs or herbal supplements known to be strong inhibitors/inducers of cytochrome P450 3A4 or cytochrome P450 2C8 within 2 weeks prior to Day 1
9. Received more than one course of radiation therapy or more than a total dose of 65 Gy. May have received radiosurgery as part of initial therapy; however, the dose counts against the total dose limit.
10. Prior taxane, vincristine, or other microtubule inhibitor chemotherapies for treatment of GBM or other malignancy
11. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
12. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
13. Any condition, including the presence of clinically significant laboratory abnormalities, which places subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study, including:

    1. Active infection including known AIDS or Hepatitis C or with a fever ≥38.5°C within 3 days prior to enrollment
    2. Diseases or conditions that obscure toxicity or dangerously alter drug metabolism
    3. Serious intercurrent medical illness (e.g., symptomatic congestive heart failure)
14. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from providing informed consent
15. Inadequately controlled hypertension (defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure > 90 mmHg)
16. Prior history of hypertensive crisis or hypertensive encephalopathy
17. New York Heart Association Grade II or greater congestive heart failure
18. History of myocardial infarction or unstable angina within 6 months prior to Day 1
19. History of stroke or transient ischemic attack within 6 months prior to Day1
20. Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
21. History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
22. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
23. Grade 2 or higher peripheral neuropathy per NCI CTCAE
24. History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
25. Serious, non-healing wound, active ulcer, or untreated bone fracture
26. Proteinuria at Screening. Subjects with a urine dipstick protein ≥2+ at Screening should undergo a 24-hour urine collection and must demonstrate ≤1g of protein in 24 hours to be eligible
27. Known hypersensitivity to inactive ingredient of bevacizumab
28. Known hypersensitivity to inactive ingredient of TPI 287
29. Pregnancy or lactation
30. Inability to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Safety of TPI 287 + bevacizumab in adults with GBM that progressed following radiation & TMZ as measured by AEs, physical/neurologic exam, KPS, weight, vital signs, hematology, serum chemistry, & urinalysis | Continuously over study treatment through 4 weeks after last dose of study drug
Phase 1: MTD of TPI 287 + bevacizumab in adults with GBM that progressed following radiation & TMZ | Within 42 days of receiving the first dose of study drug
  The MTD will be defined as the highest dose level achieved at which no more than 1 out of 6 subjects experienced a DLT that initiated within 42 days of receiving the first dose of study drug.
Phase 2: Efficacy of phase 1 MTD of TPI 287 + bevacizumab versus bevacizumab alone in adults with GBM that progressed following radiation and TMZ as measured by median PFS | Baseline & on Day 1 of each 42-day treatment cycle starting with Cycle 2, and/or as clinically indicated
  The Response Assessment in Neuro-Oncology (RANO) working group recommendations for updated response criteria for high-grade gliomas (Wen et al. 2010) will be used to determine response for this trial.

SECONDARY OUTCOMES:
Phase 1: Efficacy of TPI 287 + bevacizumab in adults with GBM that progressed following radiation and TMZ as measured by median progression free survival (PFS), overall response rate, & progression free survival rate at 4 & 6 months (PFS4 & PFS6) | Baseline & on Day 1 of each 42-day treatment cycle starting with Cycle 2, and/or as clinically indicated
Phase 2: Safety of TPI 287 + bevacizumab versus bevacizumab alone in adults with GBM that progressed following radiation & TMZ as measured by AEs, physical/neurologic exam, KPS, weight, vital signs, hematology, serum chemistry, & urinalysis | Continuously over study treatment through 4 weeks after last dose of study drug
Phase 2: Efficacy of phase 1 MTD of TPI 287 + bevacizumab versus bevacizumab alone in adults with GBM that progressed following radiation and TMZ as measured by overall survival and overall response rate | Overall response rate: baseline & on Day 1 of each 42-day treatment cycle starting with Cycle 2, and/or as clinically indicated; overall survival: up to two years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: J. P. Duic, M.D., Principal Investigator — The Long Island Brain Tumor Center at Neurological Surgery, P.C.; Samuel A. Goldlust, M.D., Principal Investigator — John Theurer Cancer Center at Hackensack University Medical Center; Louis B. Nabors, III, M.D., Principal Investigator — University of Alabama at Birmingham; Sigmund Hsu, M.D., Principal Investigator — Memorial Hermann Hospital; Nimish Mohile, M.D., Principal Investigator — University of Rochester; Tara L. Benkers, M.D., Principal Investigator — Swedish Neuroscience Institute; Jian Campian, M.D., Principal Investigator — Washington University School of Medicine; Pierre Giglio, M.D., Principal Investigator — Ohio State University
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - The Long Island Brain Tumor Center at Neurological Surgery, P.C., Commack, New York
  - The Long Island Brain Tumor Center at Neurological Surgery, P.C., Lake Success, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Memorial Hermann Hospital, Houston, Texas
  - Swedish Neuroscience Institute, Seattle, Washington